CLINICAL TRIAL: NCT06978738
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients With Relapse/Refractory Autoimmune Diseases
Brief Title: UCAR T-cell Therapy Targeting CD19/ BCMA in Patients With Relapse/ Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Lu Xuzhang, Principal Investigator, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-CE-01
Record Dates: First submitted 2025-04-28; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus; Autoimmune Hemolytic Anemia; Myasthenia Gravis; Systemic Sclerosis; ANCA-Associated Vasculitis; Inflammatory Myopathy; IgG4-RD
Keywords: Universal Allogeneic CAR T-cells; CD19/BCMA CAR T-cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anemia, Hemolytic, Autoimmune; Myasthenia Gravis; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCAR T-cell group (Experimental): A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells
  Interventions: Biological: universal allogeneic anti-CD19/BCMA CAR T-cells

INTERVENTIONS:
Biological: universal allogeneic anti-CD19/BCMA CAR T-cells — A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal allogeneic anti-CD19/BCMA CAR T-cells in With Relapse/Refractory Autoimmune Diseases.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy ofuniversal allogeneic anti-CD19/BCMA CAR T-cells in Patients With Relapse/Refractory Autoimmune Diseases.

Study intervention consists of a single infusion of universal allogeneic CART-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 years old (inclusive), regardless of gender.
* 2.Positive expression of CD19 on peripheral blood B cells confirmed by flow cytometry.
* 3.Functional requirements for major organs are as follows:

  1. Bone marrow function must meet: A. Neutrophil count ≥ 0.5×10 ^ 9/L (no colony-stimulating factor treatment within 2 weeks before examination); B. Hemoglobin ≥ 60g/L; C. Platelets ≥ 30 × 10 ^ 9/L.
  2. Liver function: Alanine aminotransferase (ALT) ≤ 3×ULN (excluding ALT elevation due to inflammatory myopathy), aspartate aminotransferase (AST)≤3×Upper limit of normal (ULN) (excluding AST elevation due to inflammatory myopathy), TBIL≤1.5×ULN (or ≤ 3.0×ULN for subjects with Gilbert syndrome);
  3. Renal function: creatinine clearance rate (CrCl) ≥ 30ml/minute (calculated by Cockcroft/Gault formula, acute CrCl decrease due to the target disease is excluded; LN is exluded);
* 4.ECOG score 0-1.
* 5.Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
* 6.Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.
* 7.Subjects with relapsed or refractory autoimmune diseases, Including relapsed or refractory Autoimmune Hemolytic Anemia, relapsed or refractory Systemic Lupus Erythematosus, relapsed or refractory or Progressive Systemic Sclerosis, relapsed or refractory or Progressive Inflammatory Myopathy, relapsed or refractory ANCA-Associated Vasculitis, relapsed or refractory Immunoglobulin-G4 related disease and relapsed or refractory Myasthenia Gravis.

Exclusion Criteria:

* 1.Subjects with a history of severe drug allergies or allergic constitutions;
* 2. Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections;
* 3. Subjects with insufficient cardiac function;
* 4. Subjects with congenital immunoglobulin deficiencies;
* 5. Subjects with a history of malignant tumors within the past five years, except for the following conditions: non-melanoma skin cancer, stage I tumors with a low recurrence probability after complete resection, clinically localized prostate cancer after treatment, cervical carcinoma in situ confirmed by biopsy or squamous intraepithelial lesion shown by smear, and stable papillary thyroid carcinoma or follicular thyroid carcinoma.
* 6. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA >ULN; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing;
* 7. Subjects with mental illness and severe cognitive dysfunction;
* 8. Pregnant women or women planning to conceive;
* 9.Subjects whom the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After UCAR T-cell Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 90 days After UCAR T-cell Infusion

SECONDARY OUTCOMES:
AIHA：Rates of CR, CRi, PR, ORR | Up to 24 Months After UCAR T-cell Infusion
  CR: complete response CRi: Complete Remission with incomplete and compensated hemolysis PR: Partial response ORR: Overall response rate
SLE：SLE Response Index 4 (SRI-4) | Up to 24 Months After UCAR T-cell Infusion
  The SRI-4 (SLE Responder Index-4) response was defined as a reduction of at least 4 points in SLEDAI score compared with the baseline level, no new British Isles Lupus Assessment Group (BILAG) A organ domain score or no more than one new BILAG B organ domain score, and no worsening in the Physician's Global Assessment (PGA) (<0.3 points worsening from the baseline level).
SLE: Change in the Systemic Lupus Erythematosus Disease Activity Index(SLEDAI) from baseline | Up to 24 Months After UCAR T-cell Infusion
  SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index, with a score of 0-6 representing mild disease activity, 7-12 representing moderate disease activity, and 12-16 representing severe disease activity
SSc：Change in the modified Rodnan Skin Score (mRSS) from baseline | Up to 24 Months After UCAR T-cell Infusion
  The modified Rodnan Skin Score (mRSS) describes the thickness of skin in 17 anatomic areas rated from 0 to 3, where 3 indicates the most severe thickening.
IIM：The ACR-EULAR Myositis Response Criteria [Total Improvement Score (TIS)] | Up to 24 Months After UCAR T-cell Infusion
  Total Improvement Score (TIS) contains Physician Global Activity(PGA)，Patient/Parent Global Activity(PtGA)，Manual Muscle Testing(MMT) and Health Assessment Questionnaire(HAQ).
  PGA:This partially validated tool measures the global evaluation by the treating physician of the overall disease activity of the patient at the time of assessment using a 10 cm. visual analogue scale and a 5 point Likert scale.
  PtGA:This partially validated tool measures the global evaluation by the patient, or by the parent if the patient is a minor, of the patient's overall disease activity at the time of assessment using a 10 cm. visual analogue scale.
  MMT:This partially validated tool assesses muscle strength using manual muscle testing (MMT). A 0 - 10 point scale is proposed for use. An abbreviated group of 8 proximal, distal, and axial muscles performs similarly to a total of 24 muscle groups, and is also proposed for use for research studies.
  HAQ:Define the health assessement questionnaire.
AAV: Change in disease activity as measured by Birmingham Vasculitis Activity Score (BVAS) | Up to 24 Months After UCAR T-cell Infusion
  The Birmingham Vasculitis Activity (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health). A negative percentage change indicated improvement in health.
IgG4-RD:IgG4-Related Disease Responder Index (IgG4-RD RI) | Up to 24 Months After UCAR T-cell Infusion
  The IgG4-RD RI detects change in disease activity and identifies improvements/worsening in the same or different organ systems. It encompasses more than 25 organs/sites and records the following for each organ/site: (i) activity trend (through a 0-3 [normal/resolved - worsening] organ/site score); (ii) presence of symptoms due to active disease; (iii) need for urgent care; (iv) presence of damage; and (v) presence of symptoms due to damage. The final activity score at each visit is obtained by summing all organ/site scores (i) and by doubling items needing urgent care (iii). Higher scores represent greater (i.e. worse) disease activity.
MG:Changes of Myasthenia Gravis Activities of Daily Living (MG-ADL) Score | Up to 24 Months After UCAR T-cell Infusion
  MG-ADL scale assesses the impact of gMG on daily functions by measuring 8 signs or symptoms that are commonly affected in MG. Each item is measured on a 4-point scale, where a score of 0 represents normal function and a score of 3 represents the loss of ability to perform that function. Total scores range from 0 to 24 points, with a higher score showing more severe MG.
MG:Quantitative Myasthenia Gravis Score (QMG) | Up to 24 Months After UCAR T-cell Infusion
  The QMG score is a 13-item scale used to quantify disease severity in myasthenia gravis. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).

CONTACTS AND LOCATIONS:
Locations (1):
- Changzhou No.2 People's Hospital, Changzhou, China

IPD SHARING:
Plan to Share IPD: No